CLINICAL TRIAL: NCT05935735
Title: Using Implementation Science to Examine the Feasibility and Efficacy of Brief Behavioral Therapy for Insomnia (BBTI) in Substance Use Disorder Recovery Programs
Brief Title: Feasibility of Brief Behavioral Therapy for Insomnia (BBTI) in SUD Recovery
Acronym: BBTI_SUDs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00343251
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Substance Use Disorders; Insomnia
Keywords: Brief Behavioral Therapy for Insomnia
MeSH Terms: conditions — Substance-Related Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BBTI Group (Experimental): Participants will receive 4 in-person sessions of Brief Behavioral Therapy for insomnia as part of their intensive outpatient treatment of substance use recovery
  Interventions: Behavioral: Brief Behavioral Therapy for Insomnia (BBTI)
- SOC Group (No Intervention): Participants will receive their usual substance abuse treatment as part of their intensive outpatient treatment of substance use recovery

INTERVENTIONS:
Behavioral: Brief Behavioral Therapy for Insomnia (BBTI) — 4 in-person sessions; 1 individual and 3 group sessions
  Arms: BBTI Group

SUMMARY:
The goal of this clinical study is to learn whether treating sleep problems is helpful in people with substance abuse problems who are living in a residential treatment program. Another goal is to study whether treating sleep problems will help individuals stay in substance abuse recovery treatment for a greater amount of time.

Participants will be asked to complete surveys at the time of enrollment and every week for the next 9 weeks for a total of 8 times. Participants will be asked to wear a watch that measures sleep (sleep watch) while the participants are in the group and for a 2-week period after the participants complete the group. Participants may also be asked to participate in an interview about the experience with the group and wearing the watch. Participants will also have "homework" throughout a 4 week period. Homework is to complete a sleep diary each morning.

The first group of 50 participants will be enrolled in the brief behavioral treatment for insomnia (BBTI) group where the participants receive typical treatment plus the sleep intervention program. The investigators will use qualitative and quantitative data to identify implementation facilitators and barriers, then further modify BBTI to improve feasibility. After modifying the BBTI protocol and re-training staff, study procedures will remain intact with the exception that the investigators will double the recruitment and randomize participants to the modified BBTI (N=50) or standard-of-care (SOC) (N=50). All participants will complete all assessments except the SOC group will not complete treatment satisfaction surveys.

DETAILED DESCRIPTION:
Brief behavioral treatment for insomnia (BBTI) is an efficacious evidence-based sleep intervention derived from cognitive behavioral therapy for insomnia (CBT-I) that may address barriers to widespread dissemination of insomnia therapy because it is brief (4 weeks), easily deliverable without need for specialty training (uses a hard-copy workbook) and behaviorally-focused. This proposal has the following two aims:

1. To use the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) framework, a well-established implementation framework that informs evaluation of health-related programs, including in community and substance use treatment settings, to evaluate the feasibility of implementing a modified BBTI among underserved special population of individuals in a residential recovery program;
2. To conduct a clinical trial to evaluate the efficacy of the modified BBTI on subjective and objective sleep outcomes compared with conventional standard-of-care. The end goal of this project is to provide empirical evidence of a modified BBTI's value in SUD recovery for individuals of diverse racial backgrounds. Successful completion of this study will promote the dissemination and sustainable adoption of an evidence-based, pragmatic, and accessible insomnia intervention in real-world SUD recovery programs.

ELIGIBILITY:
Inclusion Criteria:

* client of Cornerstone Clinic (CC); resident at Helping Up Mission (HUM)
* active SUD
* ≥ 18 years old
* ISI ≥ 8
* insomnia disorder as determined by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Sleep Disorders (SIS-D)
* able to understand English proficiently

Exclusion Criteria:

* medical or psychiatric condition interfering with treatment or requiring hospitalization
* inability to provide informed consent
* declines behavioral health treatment at CC
* suicidal ideation
* acute alcohol withdrawal requiring medical attention
* pregnant or breastfeeding
* moderate-severe sleep apnea based on WatchPAT
* restless legs syndrome based on SIS-D
* discharged from HUM

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Brief Behavioral Therapy for Insomnia (BBTI) as Assessed by the Success Rate of Outreach | Up to 1 year
  The success rate of outreach is measured by:
  * Percent of eligible Helping Up Mission (HUM) residents who were referred to study
  * Percent of eligible HUM residents who consented to study
  * Percent of HUM residents who attended BBTI Session 1
  If overall score from the three parameters above is greater than 50%, outreach is feasible
Feasibility of Brief Behavioral Therapy for Insomnia (BBTI) as Assessed by the Success Rate of Adoption | Up to 1 year
  The success rate of adoption is measured by:
  * Provider satisfaction with training as assessed by semi-structured interviews with Cornerstone Clinic researchers and staff, HUM leadership, and providers
  * Provider satisfaction with facilitating BBTI as assessed by semi-structured interviews with participants
  If overall score from the parameters above is greater than 80%, adoption is feasible
Feasibility of Brief Behavioral Therapy for Insomnia (BBTI) as Assessed by the Success Rate of Treatment Integrity | Up to 1 year
  The success rate of treatment integrity is measured by percent of maintaining treatment based on fidelity checklist.
  If overall score is above 85% treatment integrity is feasible
Changes in the Symptoms of Insomnia after Brief Behavioral Therapy for Insomnia (BBTI) as Measured by Insomnia Severity Index (ISI) | Baseline and post intervention up to 4 weeks
  Participants will complete ISI. Investigators will compare pre- and post-intervention primary outcomes. ISI is a 7-item questionnaire assessing the nature and symptoms of insomnia. ISI total score is the sum of all item scores which ranges from 0-28 and is interpreted as follows: no clinically significant insomnia (0-7), subthreshold insomnia (8-14), moderate clinical insomnia (15-21), and severe clinical insomnia (22-28). Negative changes in scores indicate improvement.
Changes in Sleep Efficiency after Brief Behavioral Therapy for Insomnia (BBTI) as Measured by Actigraphy | Baseline and post intervention up to 4 weeks
  Participants in both arms will complete daily sleep diaries and wear an actiwatch. Sleep Efficiency is a measure of total sleep time over time in bed. Higher sleep efficiency indicates improved sleep.
Changes in Substance Used Outcome as Measured by Treatment Retention [days] | Baseline and post intervention up to 4 weeks
  Treatment retention is number of days in substance used treatment. Treatment retention days will be counted by the number of days that the client is in treatment at the Helping Up Mission.

SECONDARY OUTCOMES:
Treatment Satisfaction Rate as Assessed by Treatment Satisfaction Survey | 5 Weeks
  Participants will complete a treatment satisfaction survey at the end of each BBTI session. Response options are coded from 1 to 4. The total score ranges from 5 to 20 with a higher score indicating a greater satisfaction rate.
Treatment Adherence Rate as Assessed by Treatment Adherence | 5 Weeks
  Treatment adherence is a measurement of BBTI sessions attended.
Maintenance of Intervention | Up to 1 year
  Maintenance of intervention is a measurement of treatment availability over one year.
Post-treatment Substance Use Disorder Relapse Rate as Assessed by Treatment Retention [days] | Up to 4 weeks post intervention
  Relapse Rate is percent of positive urine toxicology results. Treatment retention days will be counted by the number of days that the client is in treatment at the Helping Up Mission.
Change in Quality of life as Measured by PROMIS Global Health Scale | Baseline and post intervention up to 4 weeks
  Participants will complete the PROMIS Global Health Scale post-intervention. This is a 10-item patient-reported questionnaire that assesses healthcare-related quality of life measures. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health Score. The scores are standardized to the general population, using the "T-score" which is 50 points with a standard deviation of 10. Higher scores indicate better health.
Change in Depression Measured by PROMIS Depression Scale | Baseline and post intervention up to 4 weeks
  Participants will complete PROMIS Depression Scale questionnaires at pre-treatment and post-treatment. This is a 4-item questionnaire that assesses depressed mood in the past 7 days. The total score ranges from 8 to 40 with higher scores indicating greater severity of depression. Then, the total score is converted into T-score which is 50 points with a standard deviation of 10. Negative changes in the score indicate improvement.
Change in Anxiety Measured by PROMIS Anxiety Scale | Baseline and post intervention up to 4 weeks
  Participants will complete the PROMIS Anxiety Scale questionnaires at pre-treatment and post-treatment. This is a 4-item questionnaire that assesses the severity of the individual's anxiety in the past 7 days. The total score ranges from 7 to 35 with higher scores indicating greater severity of anxiety. Then, the total score is converted into T-score which is 50 points with a standard deviation of 10. Negative changes in the score indicate improvement.
Change in Pain Measured by PROMIS Pain Interference Scale | Baseline and post intervention up to 4 weeks
  Participants will complete the PROMIS Pain Interference questionnaire at pre-treatment and post-treatment This is a 4-item questionnaire that assesses pain interference in the last 7 days. The total score ranges from 4 to 20 with higher scores indicating greater pain interference with daily activities. Then, the total score is converted into T-score which is 50 points with a standard deviation of 10. Negative changes in the score indicate improvement.
Change in Pain Measured by PROMIS Pain Severity Scale | Baseline and post intervention up to 4 weeks
  Participants will complete the PROMIS Pain Severity questionnaire at pre-treatment and post-treatment This is a 4-item questionnaire that assesses pain intensity in the past 7 days. The total score ranges from 3 to 9 with higher scores indicating severe pain. Then, the total score is converted into T-score which is 50 points with a standard deviation of 10. Negative changes in the score indicate improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Traci J Speed, MD/PHD, Principal Investigator — Johns Hopkins University
Locations (1):
- Cornerstone at Helping Up Mission Clinic, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No